CLINICAL TRIAL: NCT00581867
Title: Intranasal Insulin and Memory in Early Alzheimer's Disease
Brief Title: Memory and Insulin in Early Alzheimer's Disease
Acronym: MAIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jeff Burns, MD (Other)
Responsible Party: Sponsor-Investigator, Jeff Burns, MD, Professor, Associate Director University of Kansas Alzheimer's Disease Center, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10896
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Insulin Aspart; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Insulin Aspart (Experimental): Participants were administered intranasal insulin aspart (40 IU) in a double-blinded fashion approximately 30 minutes prior to functional MRI scanning. After a washout period of 48 hours, participants completed the other arm. The order of saline vs. insulin was counterbalanced.
  Interventions: Drug: Insulin Aspart
- Intranasal Saline (placebo) (Active Comparator): Participants were administered intranasal saline (placebo) in a double-blinded fashion approximately 30 minutes prior to functional MRI scanning. After a washout period of 48 hours, participants completed the other arm. The order of saline vs. insulin was counterbalanced.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin Aspart — 40IU insulin aspart applied intranasally
  Other Names: intranasal insulin
  Arms: Intranasal Insulin Aspart
Drug: Placebo — Placebo
  Other Names: saline
  Arms: Intranasal Saline (placebo)

SUMMARY:
To determine which parts of the brain are involved in insulin-related memory improvement in early Alzheimer's disease and cognitively normal older adults.

DETAILED DESCRIPTION:
Functional MRI study to characterize the neuroanatomic correlates of acute exogenous insulin-related improvements in cognitive performance in early Alzheimer's disease and cognitively normal older adults. The role of the apoE-e4 allele in modulating brain insulin responses is also addressed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Early Alzheimer's disease

Exclusion Criteria:

* Patients with Late Alzheimer's disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Burns, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Hoglund Brain Imaging Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Then Intranasal Insulin: Participants in this group were randomized to receive placebo at the first fMRI visit and then received Intranasal Insulin at the second fMRI visit.
- Intranasal Insulin First, Then Placebo: Participants in this group were randomized to receive Intranasal Insulin at the first fMRI visit and then received Placebo at the second fMRI visit.
Period: First Intervention
Arm/Group | Placebo First, Then Intranasal Insulin | Intranasal Insulin First, Then Placebo
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Intranasal Insulin | Intranasal Insulin First, Then Placebo
Started | 15 (n=1 completed period 1 (placebo) but not period 2 (insulin). This individuals died between periods.) | 14 (1 individual completed period 1 (Intranasal Insulin) but did not complete period 2 (Placebo).)
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 31 total participants were enrolled in the study. 29 completed the study and had, in a counterbalanced order, one-dose of intranasal insulin followed by fMRI and over 48 hours later a dose of intranasal saline followed by fMRI.
Groups:
- Entire Study Population: Includes groups randomized to receive placebo first and insulin first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: fMRI Measure of Hippocampal Activation
Description: Percentage active voxels of total hippocampal volume of interest
Time Frame: 30 minutes After Intervention Administration
Measure: Mean (Standard Deviation); unit: percentage of active voxels
Arm/Group | Intranasal Insulin Aspart | Placebo
Number analyzed (Participants) | 29 | 29
percentage of active voxels | 36.4 (31.4) | 41.3 (33.5)

2. Secondary Outcome: Global Cognition
Description: Results derived from standardized z-score averaging performance across a battery of cognitive tests. The tests used include the Wechsler Memory Scale [WMS]-Revised Logical Memory I and II which measures a person's memory. Also used was the Wechsler Adult Intelligence Scale [WAIS] which measures intelligence in adults. The Trail Making A and B test was used to measure visual attention and task switching. The WAIS Block Design was done to test visuospatial and motor skills. The final test included in this measure is the Mini-Mental State Examination [MMSE]. The MMSE involves 30 questions and screens for cognitive impairment. Scores for each test were standardized to characterized individual global cognitive performance. The z-score reflects the standardized score. A positive z-score reflects a result above the average. A negative z-score reflects a result below the average.
Time Frame: 90 mins
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | Intranasal Insulin Aspart | Placebo
Number analyzed (Participants) | 29 | 29
z-scores | -.05 (1.15) | -.02 (1.11)

ADVERSE EVENTS:
Groups:
- Intranasal Insulin Aspart: Intranasal Insulin was administered in either first or second intervention period.
- Placebo: Placebo was administered in either first or second intervention period.
Arm/Group | Intranasal Insulin Aspart | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Insulin Aspart (N=29) | Placebo (N=29)
Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — An individual died 38 days after having one dose of intranasal saline (placebo) during the washout period due to pulmonary embolism and prior to returning for intranasal insulin. The death was considered unrelated to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes